CLINICAL TRIAL: NCT05814354
Title: A Randomized, Open, Parallel-controlled, Multicenter Phase III Trial of SHR-A1811 Versus Investigator Chemotherapy in HER2-low Expressing Recurrent/Metastatic Breast Cancer
Brief Title: SHR-A1811 Versus Investigator's Chemotherapy in Recurrent/Metastatic Breast Cancer Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-III-306
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Parallel model, randomized at a 1:1 ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- Physician's Choice (Active Comparator): Capecitabine/Eribulin/Gemcitabine/Paclitaxel/Nab-paclitaxel
  Interventions: Drug: Capecitabine/Eribulin/Gemcitabine/Paclitaxel/Nab-paclitaxel

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 is a lyophilized powder for injection intravenously. Administered according to label, as one option for Physician's Choice.
  Arms: SHR-A1811
Drug: Capecitabine/Eribulin/Gemcitabine/Paclitaxel/Nab-paclitaxel — Administered according to label, as one option for Physician's Choice (determined before randomization).
  Arms: Physician's Choice

SUMMARY:
The aim of this study was to evaluate whether the progression-free survival of SHR-A1811 was superior to investigator-selected chemotherapy in patients with HER2-low recurrent/metastatic breast cancer. To evaluate whether SHR-A1811 is superior to investigator-selected chemotherapy in patients with HER2-low recurrent/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Low-HER2 expression defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested).
2. HR-positive breast cancer with at least one endocrine therapy and disease progression was judged by the investigator to no longer benefit from endocrine therapy.
3. Has been treated with 0 to 1 prior lines of chemotherapy in the metastatic setting.
4. Has documented radiologic progression (during or after most recent treatment).
5. Has at least 1 protocol-defined measurable lesion.
6. Has protocol-defined adequate cardiac, bone marrow, renal, hepatic and blood clotting functions.
7. Fertile women (WOCBP) subjects agreed to use highly effective contraception and not to breastfeed from the time of study screening until 7 months after receiving the last study medication; a fertile woman must have a negative serum pregnancy test result within 7 days prior to the first treatment.

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable.
2. A history of human immunodeficiency virus (HIV) infection is known, or has an active autoimmune disease.
3. History of interstitial lung disease or pneumonia requiring oral or intravenous steroids.
4. Has moderate or severe cardiovascular disease.
5. Active HBV(hepatitis B) or HCV (Hepatitis C virus)-infected subjects.
6. Any other malignancies within 5 years except for those with negligible risk of metastasis or death.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Based on Blind Independent Video Review Committee (BIRC) | within approximately 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | within approximately 3 years
  Time from the date of randomization to the date of death for any cause. If there is no death reported for a participant before the data cutoff for OS analysis, OS will be censored at the last contact date at which the participant is known to be alive.
Objective Response Rate (ORR) | within approximately 2 years
  Percentage of participants who achieved a best overall response of complete response (CR) or partial response (PR), confirmed by a second assessment.
Duration of Response (DoR) | within approximately 2 years
  DoR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Clinical Benefit Rate (CBR) | within approximately 2 years
  CBR is defined as complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided